CLINICAL TRIAL: NCT02891642
Title: Liquid Biopsy With Immunomagnetic Beads Capture Technique for Malignant Cell Detection in Body Fluid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: University of California, Los Angeles (Other); M.D. Anderson Cancer Center (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Jiangsu Cancer Institute & Hospital (Other); Anhui Provincial Hospital (Other Government); Sir Run Run Shaw Hospital (Other); Renmin Hospital of Wuhan University (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: Laboratory Medicine-001
Record Dates: First submitted 2016-08-26; First posted 2016-09-07 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Malignancy; Pleural Effusion; Pleural Diseases; Ascites
Keywords: malignancy; Pleural Effusion; Pleural Neoplasms; Ascites
MeSH Terms: conditions — Neoplasms; Pleural Effusion; Pleural Diseases; Ascites; Pleural Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — body fluid for immunomagnetic separation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Malignancy, Serous effusion: Analysis of serous effusion through immunomagnetic detection device
  Interventions: Device: Immunomagnetic Detection

INTERVENTIONS:
Device: Immunomagnetic Detection — Immunomagnetic separation will be assessed through analysis of the percentage of positive samples identified compared to cytological techniques.

SUMMARY:
The purpose of the current study is to establish a Liquid biopsy method (positive enrichment by a novel immunomagnetic beads capture assay) for detection of malignant cell in serous effusions and to evaluate its sensitivity and specificity for clinical application.

DETAILED DESCRIPTION:
A serous effusion is common event in metastatic carcinoma, but it also can be associated with other benign medical conditions. Current standard method for detecting malignancy is by cytological examination. However, cytological examination is often low sensitive, often due to the large amount of fluid with relatively sparse tumor cells present and the presence of many normal cells such as mesothelial cell. The investigators have developed a new method, malignant cell enrichment with immunomagnetic beads capture followed by Pap staining and NGS, to identify target malignant cells in body fluids.

McAb NJ001 is developed for malignant cell isolation with immunomagnetic beads capture technique. This is a prospective, multi-center, double-blind, statistically powered clinical trial that will enroll patients scheduled to undergo a procedure for removal of fluid from a serous effusion with or without clinical diagnosis of caner. The purpose of the current study is to compare the novel serous effusion detection assay using NJ001 coated immunomagnetic beads capture followed by Pap staining and NGS analysis with traditional cytologic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females >18 years of age;
* Have a serous effusion;
* Scheduled for a diagnostic and/or therapeutic procedure to remove serous fluid ( Puncture of serous cavity).

Exclusion Criteria:

* Females known to be pregnant;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with serous effusion.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-09; Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Malignancies Assessed by the Liquid Biopsy with Immunomagnetic Beads Capture Technique (Cancer Cell Positive Enrichment) | The samples will be analyzed within 18 months
  SP70 positive

CONTACTS AND LOCATIONS:
Overall Officials: Shiyang Pan, MD/ PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital with Nanjing Medical University, Nanjin, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pan S, Wang F, Huang P, Xu T, Zhang L, Xu J, Li Q, Xia W, Sun R, Huang L, Peng Y, Qin X, Shu Y, Hu Z, Shen H. The study on newly developed McAb NJ001 specific to non-small cell lung cancer and its biological characteristics. PLoS One. 2012;7(3):e33009. doi: 10.1371/journal.pone.0033009. Epub 2012 Mar 30. PMID 22479355